CLINICAL TRIAL: NCT02925221
Title: Canadian Observational Cohort Study of the Real-life Assessment of Tolvaptan (JINARC™) in Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: Canadian Medical Assessment of JINARC™ Outcomes Registry
Acronym: C-MAJOR
Status: Completed | Type: Observational
Sponsor: Otsuka Canada Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 156-203-00047
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: Kidney Disease; ADPKD-Related Outcome; Quality of Life
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ADPKD patients on tolvaptan: ADPKD patients who are newly prescribed with JINARC™ (tolvaptan) or already treated with JINARC™ (tolvaptan) will be eligible.

SUMMARY:
This study is part of the Health Canada approval requirement for JINARC™ (tolvaptan) and is an observational, non-interventional study (NIS) describing the impact of tolvaptan on ADPKD-related burden of illness as measured with a set of Patient Reported Outcome (PRO) Questionnaires. The study is also describing the time to renal replacement therapy (RRT), such as dialysis and transplantation, and the long-term mortality rate and causes (i.e. renal and hepatic), in ADPKD patients treated with JINARC™ (tolvaptan)

ELIGIBILITY:
Inclusion Criteria:

* ADPKD patients ≥18 years old at the time of tolvaptan initiation
* The treating physician must have reached the decision to treat the patient with JINARC™ (tolvaptan) as per the Canadian Product Monograph prior to and independently of soliciting the patient to participate in the study
* The patient or legal guardian must have signed an informed consent indicating the understanding of the study and allowing the use of their anonymous data for the purposes of the study

Exclusion Criteria:

* The patient does not comprehend or refuses to sign the informed consent
* The patient has any contraindications to the use of JINARC™ (tolvaptan) as specified in the Canadian Product Monograph
* The patient has any condition which, as per the judgment of the treating physician, prohibits them from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adult patients newly prescribed with JINARC™ (tolvaptan) for the treatment of ADPKD, or patients who are on-treatment with JINARC™ (tolvaptan) at the time of enrolment. Investigator must be ADPKD experts qualified by experience and ability to perform the study.
Sampling Method: Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Medical Outcomes Study Short-Form 12 (MOS-SF-12v2) score | Maximum of 120 months
Changes from baseline in Autosomal Dominant Polycystic Kidney Disease-Impact Scale (ADPKD-IS) score | Maximum of 120 months
Changes from baseline in ADPKD - Pain & Discomfort Scale (ADPKD-PDS) score | Maximum of 120 months
Description of Health Care Resource Utilization | Maximum of 120 months
Work and productivity loss measured with the Work Productivity and Activity Impairment (WPAI) questionnaire | Maximum of 120 months

SECONDARY OUTCOMES:
Time to renal replacement therapy | Maximum of 120 months
Long-term mortality rate and causes | Maximum 120 months
Changes in markers of renal function | Maximum of 120 months
  Markers of renal function: Total Kidney Volume (mL); Kidney Length (cm); estimated Glomerular Filtration Rate (eGFR); Chronic Kidney Disease (CKD) stage
Adherence to treatment measured with the Medication Adherence Questionnaire | Maximum of 120 months
Time to tolvaptan treatment discontinuation | Maximum of 120 months
Long-term safety profile of tolvaptan | Maximum of 120 months
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Edmonton, Alberta
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Participants consenting to share their data are consented and identified as such in the clinical database.
Supporting Information: CSR
Time Frame: During the course of 2024, a CSR covering the study period from 2016 to the end of 2023 will be produced. Another CSR will be produced in 2026, after the conclusion of the 120-month study period.

REFERENCES:
- [Derived] McFarlane P, Bichet DG, Alam A, Bubolic S, Laplante A. Eight Years of Canadian Real-World Assessment of Tolvaptan in Patients With Autosomal Dominant Polycystic Kidney Disease: The C-MAJOR Registry. Can J Kidney Health Dis. 2026 Jan 13;13:20543581251404128. doi: 10.1177/20543581251404128. eCollection 2026. PMID 41541406